CLINICAL TRIAL: NCT07137234
Title: Efficacy of Botulinum Toxin Injection in Reducing Scar Following Cheilorrhaphy: A Randomized Controlled Clinical Trial.
Brief Title: Botulinum Toxin Injection in Reducing Scar Following Cheilorrhaphy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Basel Saeed Sayed Ahmed Shamaa, Clinical Demonstrator at oral and maxillofacial surgery department, Faculty of dentistry, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M0101025OS
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Unilateral Cleft Lip
Keywords: botulinum toxin; cleft lip; scar
MeSH Terms: conditions — Cleft Lip; Cicatrix | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I : 16 patient with unilateral cleft lip treated with surgical procedure alone (Experimental)
  Interventions: Procedure: Modified Millard rotation advancement flap technique
- Group II : 16 patients with unilateral cleft lip treated with botulinum toxin injection and surgery (Experimental)
  Interventions: Procedure: Modified Millard rotation advancement flap technique; Drug: botulinum toxin injection (BTX A) before surgical intervention

INTERVENTIONS:
Procedure: Modified Millard rotation advancement flap technique — the cleft is repaired by surgical intervention
Drug: botulinum toxin injection (BTX A) before surgical intervention — the patient will receive Botulinum toxin type A followed by surgical closure of cleft lip
  Arms: Group II : 16 patients with unilateral cleft lip treated with botulinum toxin injection and surgery

SUMMARY:
the aim of the study will be directed to evaluate clinically the effect of botulinum toxin type A injection on reducing the scar following cleft lip surgical repair.

ELIGIBILITY:
inclusion criteria :

* patients with mild to severe unilateral cleft lip requiring repair
* free from any systemic disease
* with or without cleft palate
* fit for general anesthesia exclusion criteria :
* patients with syndromic type of cleft lip
* patients with systemic disease

Min Age: 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Scar width | 3 and 6 months follow up
  Scar width will be measured by independent examiners at two at two certain points using caliper:
  point 1 (Bottom) :above the white roll. point 2 (Top): below the nasal sill.

SECONDARY OUTCOMES:
Vancouver scar scale | 3 and 6 months
  it evaluates four factors: pigmentation, pliability, height, and vascularity. it is used to asses treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Basel Saeed Shamaa, Master's, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: starting 1 year after publication